CLINICAL TRIAL: NCT06538493
Title: Jumpstarting Culturally-informed Advance Care Planning With ANAI People in Primary Care
Brief Title: Jumpstarting Advance Care Planning With ANAI People
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southcentral Foundation (Other)
Collaborators: University of Arkansas (Other); University of Washington (Other); University of Colorado, Denver (Other); Alaska Native Tribal Health Consortium (Other); University of Alaska Fairbanks (Other)
Responsible Party: Principal Investigator, Jennifer Shaw, Principal Investigator, Southcentral Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R01NR020491 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-08

CONDITIONS: Advance Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Jumpstart 1 (Experimental): Questionnaire on advance care planning experiences, preferences, and concerns
  Interventions: Behavioral: JUMPSTART-ANAI
- Jumpstart 2 (Active Comparator): Questionnaire on advance care planning experiences, preferences, and concerns plus feedback form (patient and provider)
  Interventions: Behavioral: JUMPSTART-ANAI
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: JUMPSTART-ANAI — Patient questionnaire about experiences, preferences, and concerns regarding ACP followed by feedback form with "tips" for initiating ACP conversation with provider at next clinical visit.
  Arms: Jumpstart 1; Jumpstart 2

SUMMARY:
The older Alaska Native/American Indian (ANAI) population is increasing at twice the rate of the general population with a higher burden of serious illness. Older ANAI adults with serious illness are half as likely to have advance directives (AD), indicating a need for improved access to and utilization of advance care planning (ACP) to ensure that medical care aligns with the values, goals, and preferences of ANAI patients and their families throughout the illness trajectory. The major goals of this cluster randomized trial (CRT) are to (1) evaluate the comparative effectiveness of usual care and JUMPSTART- ANAI, a culturally tailored ACP communication intervention, for prompting patient-driven ACP conversations between ANAI adults and primary care providers and to (1) identify key factors to successfully implement the intervention in health systems serving ANAI adults with serious illness.

DETAILED DESCRIPTION:
Despite a disproportionate burden of serious illness, Alaska Native and American Indian (ANAI) people are far less likely than their peers in the general US population to use palliative care, including advance care planning (ACP), which aims to align medical care with patients' values, goals, and preferences. ACP has been demonstrated to result in decreased depression, anxiety, and grief for patients and their families, increased symptom management, and fewer non-beneficial and unwanted end-of-life treatments. ACP is typically documented in advance directives (ADs) that specify patient preferences for life-sustaining treatments and who can make medical decisions on their behalf. Yet, ANAI people ages 55 and older are half as likely to have ADs as their White peers. A previous study culturally tailored and piloted an ACP communication intervention-JUMPSTART-ANAI-among 68 ANAI adults with serious illness in a Tribal health system in Alaska. This project builds on the previous study with a type 1 hybrid effectiveness-implementation trial of JUMPSTART-ANAI. The goal of this study is tailor an implementation plan for JUMPSTART-ANAI, evaluate the comparative effectiveness of the intervention and usual care for promoting patient-driven ACP communication, as measured by ADs documented in the electronic health record and identify key factors for successfully implementing JUMPSTART-ANAI in primary care systems serving ANAI adults with serious illness. Increasing access to culturally appropriate, evidence-based ACP is a high priority for Alaska Native health leaders and communities. By evaluating the effectiveness of a culturally tailored ACP intervention and tailoring implementation of the intervention for use in routine primary care, this study will generate critical information for implementing and improving palliative care services among a rapidly growing population of ANAI adults with serious illness.

ELIGIBILITY:
Inclusion Criteria:

* Alaska Native and/or American Indian
* Age 40 or older
* Empaneled to a Southcentral Foundation primary care provider
* Diagnosed with at least 1 serious illness (e.g., cancer, COPD, kidney disease)
* Has made 2 or more to primary care in last 12 months
* No Advance Directive documented in electronic health record

Exclusion Criteria:

* Cognitive impairment (≥ 2 errors) as assessed by the validated Short Portable Mental Status Questionnaire
* Not able to complete 30-minute study visit by phone or in person

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with an Advance Directive in the Electronic Health Record (EHR) | Baseline, 3 months, 6 months, 12 months
  New advance directive scanned into EHR

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Shaw, PhD, Principal Investigator — University of Alaska Fairbanks
Locations (1):
- Southcentral Foundation, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. All data owned by Tribal authority.